CLINICAL TRIAL: NCT04192188
Title: Supportive Periodontal Therapy Under Antiresorptive Therapy
Status: Completed | Type: Observational
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Dr. Antonio Ciardo, Dr. med. dent., Consultant, Heidelberg University
Other Study IDs: S-630/2019
Record Dates: First submitted 2019-12-05; First posted 2019-12-10 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Periodontitis; Antiresorptive Drugs
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ART-Group: Patients undergoing supportive periodontal therapy and independently antiresorptive therapy.
- Control Group: Patients undergoing supportive periodontal therapy without the need for antiresorptive therapy.

SUMMARY:
This observational study investigates the one-point in time and course of clinical periodontal and dental parameters during supportive periodontal therapy in patients under and without antiresorptive medication.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing supportive periodontal therapy (SPT) after completing anti-infectious therapy (AIT) in the Section of Periodontology, Clinic of Conservative Dentistry, University Hospital Heidelberg
* Regular attendance to SPT (no interruption of interval of more than one year)
* Existing radiographs (orthopantomogram or dental status) of up to six months before AIT
* ART-group: patients on antiresorptive medication (underlying diseases: osteoporosis, cancer diseases)
* Understanding of participation in this study and given informed consent

Exclusion Criteria:

* Patients < 18 years
* Patients who underwent radiation therapy
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing supportive periodontal therapy (SPT) in the Section of Periodontology, Clinic of Conservative Dentistry, University Hospital Heidelberg
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Is there a difference in the clinical attachment level between patients under antiresorptive therapy and without antiresorptive medication? | 0 months

SECONDARY OUTCOMES:
Is Intraoral digital photography suitable for DMFT and implants assessment? | 0 months
Is there a difference in the clinical attachmentlevel between baseline and 12 months after the beginning of supportive periodontal therapy in patients under antiresorptive therapy compared to patients without antiresorptive medication? | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Ciardo, Dr. med. dent., Principal Investigator — University Hospital Heidelberg
Locations (1):
- University Hospital Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Ciardo A, Simon MM, Awounvo S, Kim TS. Oral health conditions in patients under antiresorptive therapy are comparable to unexposed during supportive periodontal care. Clin Oral Investig. 2023 Nov;27(11):6523-6536. doi: 10.1007/s00784-023-05257-y. Epub 2023 Sep 15. PMID 37712984